CLINICAL TRIAL: NCT05734690
Title: COPILOT-HF: Cooperative Program for ImpLementation of Optimal Therapy in Heart Failure
Acronym: COPILOT-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Boehringer Ingelheim (Industry); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Benjamin M. Scirica, MD, Associate Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2022P002809
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Adrenergic beta-Antagonists; tocilizumab; Maximum Tolerated Dose

STUDY DESIGN:
Intervention Model Description: One group of patients, upon randomization, will immediately begin participation in a remote, pharmacist-driven heart failure clinic that will initiate and titrate medications according to a standardized medical algorithm. The comparator group will first receive curated patient education, an alert to providers, and provider education, and then after 3 months begin participation in the remote heart failure clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Medication & Education-First (Experimental): Patient will immediately begin participation in a remote, pharmacist-driven heart failure clinic that will initiate and titrate medications according to a standardized medical algorithm.
  Interventions: Drug: SGLT2i, beta blocker, ARNI, MRA, MTD
- Education-First (Active Comparator): Patient will first receive curated patient education, an alert to providers, and provider education, and then after 3 months begin participation in the remote heart failure clinic.
  Interventions: Drug: SGLT2i, beta blocker, ARNI, MRA, MTD; Behavioral: Education-First

INTERVENTIONS:
Drug: SGLT2i, beta blocker, ARNI, MRA, MTD — Immediate initiation of guideline-directed medical therapy. Will also immediately receive the same educational services provided in the "Education-First" intervention.
Behavioral: Education-First — For the first 3-months of their participation, patients in this arm will receive curated patient education, an alert to providers, provider education, and then after 3 months, be invited to participate in the remote heart failure clinic. The patient education would consist of curated video content and informational worksheets provided by email or secure patient messaging. Provider alerts would happen through notifying of a patient's eligibility for heart failure therapy. Provider education will also consist of the program's medical algorithm and a summary sheet on indications, outcomes, prescribing, and monitoring information
  Arms: Education-First

SUMMARY:
This is a randomized, open-label, initiative within the Mass General Brigham healthcare system testing two remote care strategies for optimizing the prescription of guideline-directed medical therapies in patients with heart failure, regardless of left ventricular ejection fraction (LVEF).

DETAILED DESCRIPTION:
The primary objectives are:

1. Determine if a remote, or virtual, clinic that implements a standardized, stepped-approach to guideline-directed medication optimization in patients with heart failure (across the spectrum of ejection fraction), will achieve a higher rate of guideline-directed medical therapy (GDMT) than a strategy of patient and provider education followed by remote heart failure clinic management.
2. In eligible patients with LVEF<50%, determine if the sequencing of GDMT initiation (traditional vs. sodium-glucose co-transporter-2 inhibitors-first) leads to improved GDMT intensification

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of heart failure (e.g., ICD-9 codes 428 ICD-10 codes I50 or Problem list in the electronic health record)
* Most recent EF assessed within the past 24 months
* Seen Mass General Brigham provider within the last 24 months
* English or Spanish speaking

Exclusion Criteria:

* LVEF<50% currently prescribed or intolerant to both ARNi and SGLT2i
* LVEF>50% currently prescribed or intolerant to SGLT2i
* Systolic blood pressure (SBP) <90 mmHg at last measure
* Current severe aortic stenosis or severe aortic insufficiency
* Known amyloid heart disease
* Group 1 pulmonary arterial hypertension on disease-specific therapies (e.g., Ambrisentan, Bosentan, Epoprostenol, Treprostinil, Iloprost)
* eGFR<30 mL/min/1.73m2
* Active chemotherapy
* Receiving end-of-life care or hospice
* History of transplant, currently listed above status 4 or being evaluated for transplant
* Outpatient intravenous inotrope use
* Current use of a Ventricular Assist Device
* Physician's discretion as inappropriate for remote management program

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | 3-months following randomization
  The percent of eligible enrolled patients who achieve utilization of recommended therapy for heart failure at 3 months after randomization, which includes:
  • In patients with EF<50%, utilization of 4 drug classes (ARNI/ARB/ACEI, SGLT2i, BB, and MRA),
  OR
  • In patients with EF ≥50%, utilization of SGLT2i.

SECONDARY OUTCOMES:
Secondary Endpoint | 6-months following randomization
  Any Intensification of guideline-directed medical therapy, which includes any initiation or titration of a GDMT medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blood AJ, Unlu O, Ostrominski JW, Hassan S, Nichols H, Subramaniam S, Gabovitch D, Chasse J, McPartlin M, Figueroa C, Collins E, Twining M, Varugheese M, Wagholikar K, Cannon CP, Desai AS, Scirica BM. Rationale and Design of the Cooperative Program for ImpLementation of Optimal Therapy in Heart Failure. Clin Cardiol. 2026 Feb;49(2):e70222. doi: 10.1002/clc.70222. PMID 41652651